CLINICAL TRIAL: NCT03941002
Title: Continuous Evaluation of Diaphragm Function During Assisted Mechanical Ventilation in Critically Ill Patients
Brief Title: Continuous Evaluation of Diaphragm Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, Davide Chiumello, Director of Intensive Care, University of Milan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: WOB-DiaMon
Record Dates: First submitted 2019-05-03; First posted 2019-05-07 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Respiration, Artificial; Mechanical Ventilation; Critical Illness
MeSH Terms: conditions — Respiratory Aspiration; Critical Illness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Clinical pressure support (Placebo Comparator): The level of inspiratory pressure support will be selected by the attending physician
  Interventions: Diagnostic Test: Assesment of diaphragm function
- Reduced pressure support (Active Comparator): The level of inspiratory pressure support will be reduced by 25%
  Interventions: Diagnostic Test: Assesment of diaphragm function
- Lowest pressure support (Active Comparator): The level of inspiratory pressure support will be reduced by 50%
  Interventions: Diagnostic Test: Assesment of diaphragm function

INTERVENTIONS:
Diagnostic Test: Assesment of diaphragm function — Diaphragm function will be assessed by standard mechanical parameters as assessed by esophageal and gastric pressure measurement, as well as by an ultrasonographic examination performed by an expert operator and by the continuous ultrasonographic assessment provided by the device under investigation

SUMMARY:
Aim of mechanical ventilation is to improve gas exchange and to unload the respiratory muscles delivering a form of mechanical support to the ventilation. At the same time, it is essential that the support is individually-tailored to avoid the development of muscular atrophy, a process called "ventilatory-induced diaphragm dysfunction"

Aim of the present study is that the continuous ultrasonographic assesment of diaphragm function, as obtained by the device under investigation (DiaMon, Respinor AS, Oslo, Norway) is related to the degree of effort of inspiratory muscles, as measured by gold-standard indices such as esophageal and gastric pressure measurement.

A secondary aim is that the data assessed by the device are related to a standard ultrasonographic examination performed by expert operators.

In particular, we will enroll a population of critically ill patients undergoing mechanical ventilation in assisted mode, and we will perform a decremental pressure support trial, with the following aims:

1. to evaluate the performance of a continuous and automated device for the monitoring of diaphragm contractile activity, as compared to standard mechanical indices of respiratory effort such as the pressure-time product (PTP)
2. to evaluate the performance of a continuous and automated device for the monitoring of diaphragm contractile activity, as compared to the ultrasonographic assesment of muscle function performed by an expert operator.

ELIGIBILITY:
Inclusion Criteria:

* Acute respiratory failure which necessitated endotracheal intubation and mechanical ventilation, with ventilation in pressure-support mode.
* Positive end-expiratory pressure (PEEP) lower than 10 cmH2O
* Pressure support level between 4 and 10 cmH2O
* Ratio between PaO2 and FiO2 >200 mmHg
* Resolution of the cause of respiratory failure

Exclusion Criteria:

* Diagnosis of Chronic Obstructive Pulmonary Disease (COPD)
* Pregnancy
* Circulatory failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Diaprhagm excursion | Study 1 day
  Excursion (in mm) between expiration and inspiration

SECONDARY OUTCOMES:
Esophageal pressure swing | Study 1 day
  Difference (in cmH2O) in esophageal pressure between expiration and inspiration
Pressure-time product | Study 1 day
  Integral of the area under the esophageal pressure over time (in cmH2O*sec)
Pressure-time product | Study 1 day
  Integral of the area under the trasndiaphragmatic pressure over time (in cmH2O*sec)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale San Paolo - Polo Universitario, ASST Santi Paolo e Carlo, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided